CLINICAL TRIAL: NCT03040518
Title: Feasibility Study of How Best to Engage Obese Men in Narrative SMS (Short Message System) and Incentive Interventions for Weight Loss, to Inform a Future Effectiveness and Cost-effectiveness Trial
Brief Title: Game of Stones: A Research Study That Texts Men to Help Them Lose Weight
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Stirling (Other)
Collaborators: University of Aberdeen (Other); Glasgow Caledonian University (Other); University of Glasgow (Other); University of Dundee (Other); Queen's University, Belfast (Other); University of New Brunswick (Other)
Responsible Party: Principal Investigator, Pat Hoddinott, Professor, University of Stirling
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14/185/09
Record Dates: First submitted 2016-12-16; First posted 2017-02-02 (Estimated); Last update posted 2020-04-27 (Actual); Status verified 2020-04

CONDITIONS: Obesity
Keywords: Behaviour change; Male obesity; SMS; Financial Incentive; Endowment incentive
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Narrative SMS (Experimental): Participants will receive narrative SMS for 12 months.
  Participants in all three trial arms will receive information (web or print) about weight loss and a pedometer.
  Interventions: Behavioral: Narrative SMS
- Narrative SMS and Endowment Incentive (Experimental): Participants will receive narrative SMS for 12 months. In addition, they will receive an endowment incentive for verified weight loss.
  Participants in all three trial arms will receive information (web or print) about weight loss and a pedometer.
  Interventions: Behavioral: Narrative SMS; Behavioral: Endowment Incentive
- Waiting List Control Group (No Intervention): Participants will be on a waiting list for 12 months to receive the narrative SMS which will commence after 12 month outcome data has been collected. There will be no interim measurements or contacts by the research team. Men are therefore free to choose whether to try to lose weight during the 12 months.
  Participants in all three trial arms will receive information (web or print) about weight loss and a pedometer.

INTERVENTIONS:
Behavioral: Narrative SMS — Narrative SMS have been defined as interactive life stories based around a range of characters (varying in age and socio-demographics) which can simulate the processes that make group-based interventions successful: humour, banter, peer support, facts about diet and PA and evidence based BCTs. The narrative form draws on real world learning from the film, television and games industry. When theorised, the narrative enables engagement with characters who convey the message of the intervention, and facilitate the viewer's empathy. Through creating an empathic bond with the character, users pay more attention to and become engaged and immersed within the story. This appears to lead to optimal learning and conceptualisation of the target information.
  Arms: Narrative SMS; Narrative SMS and Endowment Incentive
Behavioral: Endowment Incentive — All participants will be 'endowed' with an incentive at the start of the trial. It will be placed into a hypothetical personal account which is theirs for a year (no withdrawals). Participants will be able to secure money for verified weight loss at 3, 6, and 12 months.
  Arms: Narrative SMS and Endowment Incentive

SUMMARY:
In 2014, 24% of UK men were obese. However men rarely participate in weight loss programmes. This study looks at whether two interventions which show promise can help obese men lose weight and keep it off.

INTERVENTION 1: Sending text messages to a mobile phone. These will be written as though they come from other men who are also losing weight and include 'how to do it' diet and physical activity tips, combined with friendly humour and support.

INTERVENTION 2: The same texts plus promising men money at the start contingent on weight loss achievement. The money will vary over a year according to whether weight targets are met. This is called an endowment incentive and is based on research showing that modest payment helps people change their diet and physical activity. At the 3, 6 and 12 month weighing appointments, men will have the option of continuing with the original weight loss targets of 5%, 10% and 10% or setting lower targets of 5% of body weight at 6 months and 5% at 12 months. This is to maintain motivation and hope for men who do not meet the more ambitious weight loss targets.

This study examines if the texts work better with incentives than alone. Both interventions are delivered from a computer and have potential to reach large numbers, including men who don't use health services. This work is done together with obese men and a charity for men to help us find the best ways to deliver the interventions to as many men as possible, including men in difficult life situations.

This study will examine whether it is acceptable and feasible to randomise obese men to three groups: texts only; texts and incentive; or to a 'control group' who wait a year and then get the texts for 3 months. The feasibility of recruiting 105 obese men from two regions of Scotland will be assessed. Half of the men will get an invitation letter from their GP. The other half will be approached in the community, given information about the study and invited to take part. Men can take part if their waist circumference is 40 inches and more or their Body Mass Index is 30 or higher. The study examines how long it takes to find 105 obese men who want to take part, how many come back to suitable venues at 3, 6 and 12 months to get weighed and answer questions about their quality of life, lifestyle and motivation. At the end participants will report about their experiences of weight loss and of being in the study.

ELIGIBILITY:
Inclusion Criteria:

* Obese adult men aged 18 or over with and without known health conditions, who do or do not access GP services. Obesity is defined as a BMI equal to or over 30 and/or a waist circumference measurement equal to or above 40 inches (102cm)

Exclusion Criteria:

* Insufficient English language for SMS intervention; no mobile phone access.
* Planning to move out of the area within 12 months.
* Current or recent participation in a research weight loss intervention study (in the last 3 months).
* For GP recruitment: severe medical, terminal or psychiatric illness (patient or close family member)
* Impaired cognitive function that would limit understanding of study information and SMS messages.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2019-11-30 (Actual)

PRIMARY OUTCOMES:
Decision whether to proceed to full RCT (Composite Measure) | 12 months
  A decision whether to proceed to a full effectiveness and cost-effectiveness RCT for the SMS intervention, with or without an incentive, compared to a waiting list control. This will be based on the progression criteria:
  1. Acceptability of the intervention and the control group (willingness to be randomised, intervention engagement, participant retention, qualitative views)
  2. Feasibility of recruiting 105 men in 4 months
  3. 12 month outcomes on at least 72 % of men randomised per group
  4. Evidence of mean weight loss of at least 3% of baseline weight at 12 months in any intervention group
  An Independent Trial Steering Committee will decide whether the findings support a two or three arm trial or not

SECONDARY OUTCOMES:
Weight | 3, 6 and 12 months
BMI | 3, 6 and 12 months
Waist circumference | 3, 6 and 12 months
Fruit and vegetable consumption | 6 and 12 months
  "How many portions of fruit and vegetables (including pulses, salad, vegetables, fruit juices and fresh, dried and canned fruit) did you eat yesterday?" Answered on a scale of none to 7 or more
Physical activity | 6 and 12 months
  International Physical Activity Questionnaire items:
  'During the last 7 days, on how many days do you do moderate physical activities like carrying light loads, bicycling at a regular pace or walking?' Answered on a scale of days per week (none to 7) 'During the last 7 days, how much time did you spend sitting?' On a week day? (Answered in hours and minutes) On a weekend day? (Answered in hours and minutes)
Smoking status | 6 and 12 months
  'Do you currently smoke or have you ever smoked?' Choose from; Yes, I currently smoke every day; Yes, I currently smoke, but not every day; Yes, I used to smoke but have quit or No, I have never smoked.
Alcohol consumption | 6 and 12 months
  'During the last month, how many days did you usually have any kind of drink containing alcohol?' Choose from: Everyday; 5 to 6 times a week; 3 to 4 times a week; twice a week; once a week; 2 to 3 times a month; once a month or never
EQ-5D-5L | 6 and 12 months
  EQ-5D-5L
Health Service Use | 6 and 12 months
  Over the LAST 3 MONTHS, have you used any of the following NHS Services? Choose from: Your GP or another GP Nurse Doctor or nurse in an emergency department (causality/ A&E) Outpatient appointments Inpatient stay
  Yes/No
Wellbeing | 12 months
  Warwick and Edinburgh wellbeing questionnaire

OTHER OUTCOMES:
Confidence in weight loss and weight loss maintenance | 3, 6 and 12 months
  'How confident are you in your ability to lose weight? Scale from 1 (not confident) to 7 (very confident). 'How confident are you in your ability to keep lost weight off in the long term? Scale from 1 (not confident) to 7 (very confident).
Importance of weight loss | 3, 6 and 12 months
  'How important is losing weight for you at the moment?' Scale from 1 (not important) to 7 (very important).
Weight loss maintenance perceptions | 3, 6 and 12 months
  The below questions ask you about your weight loss in the last 3 months Items Items below rated strongly disagree, disagree, agree or strongly agree.
  In the last 3 months; I was; motivated to lose weight; tired most of the time; stressed most of the time; hungry most of the time; having to think a lot about my weight loss plan; following my weight loss plan without having to think much about it; satisfied with the results of my weight loss; enjoyed following my weight loss plan; doing things which conflicted with my weight loss plan; doing things which helped me with my weight loss plan; supported by my friends and family to stick to my weight loss plan; in places and situations that made it difficult to follow my weight loss plan.
Weight loss techniques | 3, 6 and 12 months
  Have you done any of the following over the last 3 months?' Choose from; not at all; 1-2 times a month; about weekly or every day or most days.
  Tried to limit what you eat or drink to try to lose weight?; done an exercise workout (including video/ DVD workouts) at home?; attended a commercial weight loss programme (e.g. Weight Watchers); attended a gym, leisure centre or local sport facility to swim or take part in other psychical activity sessions?, attended a weight-reduction clinic at your GP surgery or another NHS setting?
Weight maintenance focus | 3, 6 and 12 months
  If my weight stays the same for the next 3 months I would consider it a success, even if I don't lose any If my weight stays the same for the next 3 months I would be happy, even if I don't lose any. Scale from 1 (strongly disagree) to 7 (strongly agree).
  'I am trying to maintain my weight loss at the moment rather than trying to lose more weight' Scale from 1 (strongly disagree) to 7 (strongly agree).
Automaticity | 3, 6 and 12 months
  'Eating fruits and vegetables is something I do automatically' Scale from 1 (strongly disagree) to 7 (strongly agree) 'Being psychically active is something I do automatically' Scale from 1 (strongly disagree) to 7 (strongly agree)
Self-regulation of eating behaviour | 3, 6 and 12 months
  Self-Regulation of Eating Behaviour Questionnaire (SREBQ - Kliemann et all., 2016; doi: 10.1186/s12966-016-0414-6)

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - NHS Greater Glasgow and Clyde, Glasgow
  - NHS Forth Valley, Stirling

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] McDonald MD, Dombrowski SU, Skinner R, Calveley E, Carroll P, Elders A, Gray CM, Grindle M, Harris FM, Jones C, Hoddinott P; Game of Stones team. Recruiting men from across the socioeconomic spectrum via GP registers and community outreach to a weight management feasibility randomised controlled trial. BMC Med Res Methodol. 2020 Oct 6;20(1):249. doi: 10.1186/s12874-020-01136-2. PMID 33023501
- [Derived] Dombrowski SU, McDonald M, van der Pol M, Grindle M, Avenell A, Carroll P, Calveley E, Elders A, Glennie N, Gray CM, Harris FM, Hapca A, Jones C, Kee F, McKinley MC, Skinner R, Tod M, Hoddinott P. Game of Stones: feasibility randomised controlled trial of how to engage men with obesity in text message and incentive interventions for weight loss. BMJ Open. 2020 Feb 25;10(2):e032653. doi: 10.1136/bmjopen-2019-032653. PMID 32102807
- See also: Main results paper in BMJ Open — https://bmjopen.bmj.com/content/bmjopen/10/2/e032653.full.pdf